CLINICAL TRIAL: NCT04519216
Title: Breastfeeding Education in the Time of COVID-19. Hybrid Telesimulation With Standardized Patients for Pediatric and Family Medicine Trainees, a Randomized Trial
Brief Title: Breastfeeding Education in the Time of COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1613611
Record Dates: First submitted 2020-08-12; First posted 2020-08-19 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Breastfeeding; Breastfeeding, Exclusive; Breastfeeding Jaundice; Educational Problems
MeSH Terms: conditions — Breast Feeding; Breastfeeding Jaundice

STUDY DESIGN:
Intervention Model Description: This is a prospective cluster randomized controlled trial of a novel educational intervention in pediatric and family medicine residents during the nursery rotation. In this study, we will enroll 1st year pediatric and family medicine residents and 3rd year supervising pediatric residents on their newborn nursery 4-week rotation and randomization will occur clustered by rotation month. The educational intervention will be conducted during the first week of the rotation. Both groups will complete pre-intervention survey that collects demographic information, personal infant feeding experiences, and any breastfeeding medicine experience. All participants will be invited to complete a free online course (Lactation Support in a Telehealth Setting Course) prior to the telemedicine intervention or control group discussion with the clinical pediatrician.
Who Masked: Outcomes Assessor
Masking Description: Outcomes are blinded to the assessor when completing the trial data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional education (Active Comparator): Participants in the control group will complete an online unfolding case scenario. Then these same participants will participate in a videoconferencing case based lecture with the academic pediatric fellow
  Interventions: Behavioral: Telesimulation
- Telesimulation (Experimental): Participants in the intervention group will complete an online unfolding case scenario. Then these participants will complete a telesimulation case with a standardized patient via video conferencing.
  Interventions: Behavioral: Telesimulation

INTERVENTIONS:
Behavioral: Telesimulation — Telesimulation educational intervention

SUMMARY:
This project will establish that pediatric and family medicine residents who complete a hybrid breastfeeding medicine curriculum that includes an asynchronous unfolding case scenario along with telesimulation with a standardized patient (SP) will provide timely, skilled lactation support more frequently than residents randomized to an asynchronous unfolding case scenario followed by videoconference group discussion regarding care for the breastfeeding dyad.

DETAILED DESCRIPTION:
1. Establish that pediatric and family medicine residents who complete a novel breastfeeding medicine curriculum that includes an online unfolding case scenario along with telemedicine simulation with a standardized patient (SP) will provide timely, skilled lactation support more frequently than residents randomized to an online unfolding case scenario followed by traditional didactic breastfeeding case-presentation via videoconference.
2. Establish that online learning via unfolding case scenario and telemedicine simulation with a SP will be feasible for family medicine and pediatric residents to complete during their newborn nursery rotation.

Intern and third year residents completing their newborn nursery rotation at UC Davis Medical Center will be cluster-randomized by rotation month to receipt of breastfeeding education via telesimulation with standardized patient or traditional case-based learning via videoconferencing with pediatric faculty. The primary outcome of this study will be the translation of clinical lactation skills to the care of breastfeeding mothers and newborns. I hypothesize that pediatric and family medicine residents randomized to complete the telesimulation with SP will translate their acquired clinical lactation skills to the care of breastfeeding mothers and newborns at a greater rate than residents who complete a videoconference case-based traditional curriculum discussion with a newborn nursery pediatrician.

ELIGIBILITY:
1. Inclusion Criteria: Pediatric and Family Medicine resident physicians at UC Davis Medical Center
2. Exclusion criteria: Individuals who are unable to communicate in English, Individuals who do not have access to videoconferencing via computer or phone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Change in practice patterns | at enrollment, 2 weeks and 3 months following intervention
  Breastfeeding medicine practice patterns of physician residents will be assessed at enrollment and following the intervention/control. Physician resident participants will complete a survey querying the number of times they have counseled patients about breastfeeding, the number of breast examinations performed, the number of witnessed breastfeeding sessions, and any experience with counseling about manual expression of breast milk.

SECONDARY OUTCOMES:
Self efficacy | at enrollment, 2 weeks and 3 months following intervention
  Physician residents (participants) will fill out a survey about their breastfeeding counseling self efficacy prior to and after the intervention.
Satisfaction with simulation | Immediately following the educational intervention
  Physician residents (participants) will fill out a survey about their satisfaction with the breast feeding medicine curriculum after the educational intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Hoyt-Austin, DO, Principal Investigator — University of California, Davis
Locations (1):
- University of California - Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No